CLINICAL TRIAL: NCT00602914
Title: An Open Label Study in Healthy Volunteers and Diabetes Mellitus Type II Subjects to Determine the Safety, Pharmacokinetics and Pharmacodynamics Profile of Insulin Injected by the MicronJet Device
Brief Title: A Pilot Study to Assess the Safety, PK and PD of Insulin Injected Via MicronJet or Conventional Needle
Acronym: MicronJet
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NP-1-001
Record Dates: First submitted 2007-12-30; First posted 2008-01-28 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2008-04

CONDITIONS: Intradermal Injections
Keywords: MicronJet (microneedles); Intradermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 10 healthy volunteers will receive 0.1 U/kg. Once administered with a conventional needle (SQ) and then with MicronJet needle (ID) in a randomized order
  Interventions: Device: MicronJet
- 2 (Experimental): 10 Type II DM subject will receive 0.2 U/kg. Once administered with a conventional needle (SQ) and then with MicronJet needle (ID) in a randomized order
  Interventions: Device: MicronJet

INTERVENTIONS:
Device: MicronJet — The micronJet is a microneedle injection device designed for intradermal delivery of drugs (i.e. delivery into the skin). In this study the MicronJet will be used to inject insulin vs. a convention needle injection.
Device: MicronJet — MicronJet, Intradermal Injection
  Other Names: Microneedles

SUMMARY:
The purpose of this study is to compare glucose pharmacokinetics and insulin pharmacodynamics injected via the MicronJet in comparison with a conventional needle.

DETAILED DESCRIPTION:
Administration of insulin to the skin has many potential advantages including improved kinetics and reduced pain. Today, insulin is injected to the SQ space, using, in most cases, various devices incorporating standard metal needles and usually causing considerable pain and discomfort to the patients. NanoPass has developed a microneedle based needle substitute for intradermal injections. This device requires minimal expertise and is expected to cause minimal or no pain during injections.

The objective of this study is to compare the pharmacokinetics and pharmacodynamics of insulin Novorapid® (Novo Nordisk) injected via the MicronJet device intradermally, to a conventional needle injected to the SQ space.

ELIGIBILITY:
A. Healthy volunteers

Inclusion Criteria:

1. Men ranging in age from 18-40 years.
2. In good general health as determined by medical history, physical examination, ECG and clinical laboratory tests obtained with 14 days prior to the start of the study.
3. BMI<30 or the volunteer is not considered obese by the Principal Investigator with a written statement at screening.
4. Willing and able to abide by the dietary requirements of the study.
5. Willing and able to give written informed consent in a manner approved by the Institutional Review Board or Ethics Committee.

Exclusion Criteria:

1. History of known or suspected clinically significant hypersensitivity to any drug.
2. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Clinically significant cardiovascular, hepatic, gastrointestinal, metabolic, neurological, pulmonary, endocrine, psychiatric, coagulation or neoplastic disorders.
4. Participation in radiologic studies involving parenteral administration of iodinated contrast materials within two weeks prior to screening.
5. Subjects with history of recent alcohol abuse (defined as consumption of more than 21- ml of alcohol per week; or the equivalent of fourteen 4-oz glasses of wine, fourteen 12 oz can/bottle of beer or wine cooler) or other substance abuse.
6. Any protocol-required laboratory test abnormality that is considered clinically significant.
7. Participation in another investigational drug study within 90 days before the first day of dosing.
8. History of non-compliance to medical regimens, or subjects who are considered potentially unreliable.
9. Blood or plasma donation within the past 90 days.
10. Mentally unstable or incompetent.
11. Positive hepatitis C screen or positive hepatitis B screen.
12. HIV positive

B. Type 2 diabetic patients

Inclusion Criteria:

1. Type 2 male patients and post-menopausal females aged 30-70 years.
2. HA1c 6.5-10%
3. Naïve or treated with Metformin only
4. BMI< 35
5. Willing and able to abide by the dietary requirements of the study.
6. Willing and able to give written informed consent in a manner approved by the Institutional Review Board or Ethics Committee.

Exclusion Criteria:

1. History of known or suspected clinically significant hypersensitivity to any drug.
2. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Clinically significant cardiovascular, hepatic, gastrointestinal, metabolic, neurological, pulmonary, endocrine, psychiatric, coagulation or neoplastic disorders.
4. Participation in radiologic studies involving parenteral administration of iodinated contrast materials within two weeks prior to screening.
5. Subjects with history of recent alcohol abuse (defined as consumption of more than 21- ml of alcohol per week; or the equivalent of fourteen 4-oz glasses of wine, fourteen 12 oz can/bottle of beer or wine cooler) or other substance abuse.
6. Any protocol-required laboratory test abnormality that is considered clinically significant.
7. Participation in another investigational drug study within 90 days before the first day of dosing.
8. History of non-compliance to medical regimens, or subjects who are considered potentially unreliable.
9. Blood or plasma donation within the past 90 days.
10. Mentally unstable or incompetent.
11. Positive hepatitis C screen or positive hepatitis B screen.
12. HIV positive

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Blood samples for PK and PD will be collected | pre dose and up to 360 minutes post dose of administration

SECONDARY OUTCOMES:
Feedback from study participants and staff on their overall impression with the MicronJet device, using questionnaires | All study duration

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Head, Diabetes Unit, Hadassah Medical Organization, Jerusalem, Israel